CLINICAL TRIAL: NCT05128721
Title: A Phase 1 Clinical Trial to Evaluate the Safety, Tolerability, and Immunogenicity of Inactivated Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2) Vaccine Against COVID-19 in Healthy Adults
Brief Title: Evaluation of Inactivated Vaccine in Healthy Adults Against Coronavirus Disease of 2019 (COVID-19)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Research Centre, Egypt (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NO-B041
Record Dates: First submitted 2021-11-12; First posted 2021-11-22 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: COVID-19; Vaccine Reaction; Vaccine Adverse Reaction
Keywords: COVID-19; Inactivated SARS-CoV-2 Vaccine; NRC-VACC-101; Vaccine Safety; Vaccine Tolerability; Vaccine Immunogenicity; Covi Vax; Egyptian Inactivated SARS-CoV-2 Vaccine
MeSH Terms: conditions — COVID-19 | interventions — NRC-VACC-101 vaccine

STUDY DESIGN:
Intervention Model Description: A Randomized, Open-label, Phase 1 Clinical trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NRC-VACC-101 vaccine 3 microgram (Active Comparator): Volunteers will receive two IM doses of the vaccine, concentrations of 3 mcg, 28 days apart.
  Interventions: Biological: Covi Vax
- NRC-VACC-101 vaccine 6 microgram (Active Comparator): Volunteers will receive two IM doses of the vaccine, concentrations of 6 mcg, 28 days apart.
  Interventions: Biological: Covi Vax
- Control arm (Placebo Comparator): Volunteers will receive two IM doses of the placebo (excipients only), 28 days apart.
  Interventions: Biological: Covi Vax

INTERVENTIONS:
Biological: Covi Vax — Inactivated SARS-COV-2 Vaccine/alum adjuvant preparation in addition to excipients (NRC-VACC- 101) administered as an IM Injection. NRC-VACC-101 is provided as a single dose of inactivated vaccine of opaque white liquid free from visible particles filled in injection vial (2R) glass vials. Each Dose of Covi Vax Vaccine contains 6 mcg antigen of A human coronavirus (hCoV)-19/Egypt/NRC-03/2020 SARS-CoV-2 strain.
  Other Names: NRC-VACC-101 vaccine; Egyptian Inactivated SARS-CoV-2 Vaccine; NRC Inactivated SARS-CoV-2 Vaccine

SUMMARY:
In this phase 1 study, the inactivated virus vaccine National Research Centre (NRC) Vaccine-101 (VACC-101) will be investigated for its safety and immunogenicity in healthy volunteers with the aim of providing effective and safe protection against COVID-19.

DETAILED DESCRIPTION:
This is a Phase I, Randomized, Open-Labeled Clinical trial. Eligible volunteers will be randomized in a 1:1:1 allocation ratio, into one of the three study arms using the Interactive Web Response Technology (IWRS).

Unscheduled visits can occur at any time during the study period outside the initially planned study visits, all the extra visits will be documented in the subjects' files. Volunteers will be randomized into one of the following arms to receive different doses of the Inactivated

SARS-COV-2 Vaccine "NRC-VACC-101" as an intramuscular (IM) Injection or Placebo:

Arm One:

Volunteers will receive two IM doses of the vaccine, concentrations of 3 mcg, 28 days apart.

Arm Two:

Volunteers will receive two IM doses of the vaccine, concentrations of 6 mcg, 28 days apart.

Arm Three (Control arm):

Volunteers will receive two IM doses of the placebo, 28 days apart. The first 9 subjects will be initially vaccinated with their first dose, as per their assigned study arm determined by the randomization procedures and will be followed up until day 14 (visit 03). At this point in the study, the Data Safety and Monitoring Board (DSMB) will review safety data before proceeding with vaccinating the rest of the recruited subjects

ELIGIBILITY:
Inclusion Criteria:

1. Adults with age 18 to 50 years.
2. Willingness.
3. For married females of childbearing age: Willingness to practice continuous effective contraception for one year from the start of the study.
4. Agreement to refrain from blood donation during the study.
5. Body temperature is within the normal range (36.5 - 37.5°C).
6. General good health as established by medical history, physical and laboratory examinations.

Exclusion Criteria:

1. Pregnancy or lactation.
2. Inability to provide informed consent.
3. Recent receipt of any vaccination within 30 days prior to baseline.
4. Planning to receive any vaccination during the course of the study.
5. Prior receipt of Adenovirus vaccine, or any other Coronavirus vaccine.
6. Recent receipt of any immunoglobulin within 90 days prior to baseline.
7. Recent receipt of any blood product within 90 days prior to baseline.
8. Volunteers who are immunosuppressed or receiving immunosuppressive medications, including:

   HIV infection, asplenia, recurrent severe infections, and the use of immunosuppressive medications within the past 6 months, except for topical steroids or short-term oral steroids (course lasting < 14 days).
9. Currently taking any product (investigational or off-label) for prevention of COVID-19 disease.
10. Having any autoimmune disease.
11. History of allergic reactions for any of the vaccine components.
12. History of angioedema.
13. History of anaphylaxis.
14. History of cancer.
15. History of serious psychiatric conditions that are likely to affect participation in the study.
16. Having bleeding disorders.
17. Having chronic respiratory diseases.
18. Having chronic cardiovascular disease, gastrointestinal disease, liver disease, renal disease, endocrine disorders, and neurological illness.
19. Volunteers with BMI ≥ 40 Kg/m2 or ≤ 18 Kg/m2.
20. Current alcohol abuse.
21. Drug abuse within 5 years prior to baseline.
22. History of laboratory-confirmed COVID-19 or seropositivity for SARS-CoV-2 or positive serum immunoglobulin M (IgM) and immunoglobulin G (IgG) to the SARS CoV-2 or abnormal chest CT-Scan (COVID-19 image) or positive pharyngeal/sputum swabs for SARS-CoV-2.
23. Participation in other studies involving study intervention within 28 days prior to study entry and/or during study participation.
24. High-risk population (volunteers who work in front-line health facilities or were in close contact with confirmed COVID-19 cases).
25. Living in the same household as anyone at high risk of severe COVID-19.
26. Any condition, according to the judgment of the investigator, that would interfere with the subject's ability to comply with all study requirements or that would place the subject at unacceptable risk by his/her participation in the study or impair the interpretation of the study data.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-11-14 (Actual); Primary Completion 2023-02-23 (Estimated); Study Completion 2023-05-23 (Estimated)

PRIMARY OUTCOMES:
The safety of NRC-VACC-101 Vaccine | Follow up for any solicited adverse event(AE) reported within 7 days
  To evaluate the safety of the proposed regimens of NRC-VACC-101
The tolerability of NRC-VACC-101 Vaccine | Follow up for any AE within 28 days of each dose
  To evaluate the tolerability of the proposed regimens of NRC-VACC-101 Vaccine in the healthy population

SECONDARY OUTCOMES:
The seroconversion rate of neutralizing antibodies | The evaluation of the antibody will be measured up to one month of each dose
  To evaluate the seroconversion rate of neutralizing antibodies resulting from the NRC-VACC-101 Vaccine
To recommend the dose level of NRC-VACC-101 Vaccine for the phase II trial. | The evaluation of the Microneutralization Assay will be assessed up to one month of each dose
  The evaluation of the Microneutralization Assay curve will give an overview of the dose possible suggested dose of NRC-VACC-101 Vaccine for the phase II trial

CONTACTS AND LOCATIONS:
Overall Officials: Osama Azmy, MD, Principal Investigator — Medical Research and Clinical Studies Institute National Research Centre, Dokki, Giza, Egypt.
Locations (1):
- Medical Research Centre of Excellence National Research Centre, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon individual request.
Supporting Information: Study Protocol, ICF
Time Frame: About one year after completion of the trial
Access Criteria: Data will be shared upon individual request by contacting the sponsor of the trial.